CLINICAL TRIAL: NCT05811169
Title: Quest for Tumour Evolution of Non-small Cell Lung Cancer in Chinese (Unicorn-Quest)
Brief Title: Quest for Tumour Evolution of Non-small Cell Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Queen Elizabeth Hospital, Hong Kong (Other); Pamela Youde Nethersole Eastern Hospital (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other); Princess Margaret Hospital, Hong Kong (Other Government); Tuen Mun Hospital (Other Government); United Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UW 20-145
Record Dates: First submitted 2023-02-26; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Next Generation Sequencing
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The formalin-fixed paraffin embedded tumour and lymph node samples of non-small cell lung cancer as well as blood, plasma and serum samples are retrieved and collected for next-generation sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Early or metastatic non-small cell lung cancer: The formalin-fixed paraffin-embedded specimen will be retrieved for next generation sequencing.
  Interventions: Genetic: Next generation sequencing

INTERVENTIONS:
Genetic: Next generation sequencing — Next generation sequencing

SUMMARY:
To study and comprehend the evolutionary and genomic landscape between primary and metastatic sites and the dynamics of intratumour and intertumour heterogeneity over time with reference to the treatment modalities for each Chinese patient with non-small cell lung cancer.

DETAILED DESCRIPTION:
The importance of intratumour and intertumour heterogeneity in non-small cell lung cancer has been extensively interrogated recently. However there is a lack of similar data associated with treatment and survival outcomes in Chinese population. Unicorn-Quest, a prospective observational study of Chinese patients with either primary or metastatic non-small cell lung cancer, aims to identify the evolutionary changes from the primary tumour, regional nodes and distant metastases of the same patients and among different patients, through multiregion and longitudinal tumour and nodal collection with next-generation sequencing. By following non-small cell lung cancer from early stage to relapse or distant metastasis, identifying the changes of genomic landscape with correlation with treatment and survival outcomes, this study may help identify unique cancer trajectories and novel therapeutic targets for non-small cell lung cancer in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent
* Patients ≥18 years of age, with histologically confirmed non-squamous non-small cell lung cancer who plan to receive active anti-cancer treatment for their non-small cell lung cancer.
* Sufficient tissues with a minimum of two tumour or nodal regions are available for the study based on pre-operative imaging and post-operative pathological findings.

Exclusion Criteria:

* Any other* malignancy diagnosed or relapsed at any time, which is currently being treated (including by hormonal therapy).

Any other* current malignancy or malignancy diagnosed or relapsed within the past 3 years**.

*Exceptions are: non-melanomatous skin cancer, stage 0 melanoma in situ, and in situ cervical cancer

**An exception will be made for malignancies diagnosed or relapsed more than 2, but less than 3, years ago only if a pre-operative biopsy of the lung lesion has confirmed a diagnosis of NSCLC.

* Psychological condition that would preclude informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stage I to IVB non-squamous non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intratumour heterogeneity | 5 years
  Number of participants who have single actionable and non-actionable genetic mutations and multiple actionable and non-actionable genetic mutations within the same groups of patients with early and metastatic non-small cell lung cancer
Intertumour heterogeneity | 5 years
  Number of participants who have single actionable and non-actionable genetic mutations and multiple actionable and non-actionable genetic mutations of different groups of patients with early and metastatic non-small cell lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Victor Ho-Fun Lee, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No